CLINICAL TRIAL: NCT06063070
Title: An Open, Multicenter, Exploratory Clinical Study of Fluzoparib in Combination With Bevacizumab for Maintenance Therapy After First-line Platinum-containing Chemotherapy in BRCA Wild-type Advanced Ovarian Cancer
Brief Title: First-line Maintenance Treatment With Fluzoparib Plus Bevacizumab in Advanced BRCA Wild Type Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-321-01
Record Dates: First submitted 2023-09-19; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer; High Grade Serous Adenocarcinoma of Ovary; High Grade Endometrioid Ovarian Cancer; Primary Peritoneal Cancer; Fallopian-tube Cancer
Keywords: ovarian cancer; PARP inhibitors; Flzuoparib; Antiangiogenic agents; Bevacizumab; BRCA wild-type
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — fluzoparib; Poly A; Adenosine Diphosphate Ribose; Bevacizumab; Angiogenesis Inhibitors

STUDY DESIGN:
Intervention Model Description: Drug: fluzoparib plus Bevacizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib + Bevacizumab (Experimental): Fluzoparib capsule: oral administration, 3 capsules/dose (150 mg/ dose), twice a day, in the morning and evening, before/after meals can be taken orally, it is recommended to take orally within 0.5h after breakfast and dinner, continuous administration. Every 3 weeks is a treatment cycle.
  Bevacizumab injection: intravenous, 15 mg/kg, every 3 weeks for a treatment cycle until disease progression or intolerable toxicity, up to a total of 15 months.
  Interventions: Drug: Fluzoparib Capsules; Drug: Bevacizumab

INTERVENTIONS:
Drug: Fluzoparib Capsules — oral
  Other Names: Poly (ADP-ribose) polymerase (PARP) inhibitor
Drug: Bevacizumab — Injectable solution
  Other Names: Antiangiogenic agents

SUMMARY:
This is an open-label, multi-center Phase II study of fluzoparib combined with bevacizumab for maintenance therapy after first-line platinum-containing chemotherapy in patients with BRCA wild-type advanced ovarian cancer. The primary objective is to evaluate median progression free survival of fluzoparib plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and ability to comply with treatment and follow-up.
2. Age ≥ 18 years (Calculated on the date the informed consent was signed).
3. Pathologically confirmed high-grade serous (or medium-low differentiation) or high grade endometrioid (≥ grade II) ovarian cancer, primary peritoneal cancer and/or fallopian-tube cancer:

   - Mixed tumors: high-grade serous or high grade endometrioid (≥ grade II) component must be >50%.
4. Patients with newly diagnosed, histologically confirmed, advanced (FIGO stage III or IV of the 2018 FIGO classification) ovarian, fallopian tube, or primary peritoneal cancer; and underwent tumor reduction surgery.
5. Patients must have received prior to enrollment a minimum of 6 cycles and a maximum of 9 cycles of first line platinum-taxane chemotherapy. However, if platinum-based therapy must be discontinued early as a result of intolerable toxicity, patients must have received a minimum of 4 cycles of the platinum regimen:

   -Preoperative neoadjuvant chemotherapy and postoperative chemotherapy counted as 1 chemotherapy treatment regimen.
6. Patients must be prior to enrollment in complete response (CR) or partial response (PR) from their first line treatment, and use of the trial drug at least 3 weeks and no more than 9 weeks after their last dose of chemotherapy.

   * At least 4 cycles of the platinum regimen treatment were completed.
   * During or after platinum-containing chemotherapy, concurrent use of other investigational drugs and treatment other than endocrine therapy drugs are not permitted.
   * Bevacizumab in combination with the first line platinum-taxane chemotherapy was allowed.
   * At the end of the last platinum-containing regimen, the radiographic evaluation of the efficacy was CR or PR, CA125 was reduced to within the upper limit of normal (ULN) or ≥90% lower than pre-treatment levels during treatment, and CA125 was maintained at <1x ULN or has not >10% higher than previously observed for 7 days before the first trial of drug administration.
   * If there is no evaluable lesion prior to chemotherapy, CA125 must remit to <Upper Limit of Normal (ULN) during treatment and CA125 should be maintained at <1x ULN for 7 days prior to the first trial dose.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. Germline BRCA1/2 wild-type.
9. Patients must have normal organ and bone marrow function (use of any blood components and cell growth factors within 14d prior to the first dose is not permitted):

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
   2. Platelets count ≥ 100 x 109/L;
   3. Hemoglobin ≥ 9 g/dL;
   4. Serum albumin ≥ 3 g/dL;
   5. Bilirubin ≤ 1.5x ULN;
   6. Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN;
   7. Serum creatinine ≤ 1.5x ULN;
10. Postmenopausal or evidence of non-childbearing status for women of childbearing potential prior to the first dose of study treatment.

Exclusion Criteria:

1. Previous (within 5 years) or concurrent with other uncured malignant tumors, except for cured skin basal cell carcinoma, cervical carcinoma in situ and breast cancer with no recurrence >3 years after radical surgery;
2. Patients with untreated central nervous system metastases:

   -Patients with prior treatment (radiotherapy or surgery) for systemic, radical brain or meningeal metastases may be enrolled if imaging confirms that stabilization has been maintained for at least 1 month and systemic hormone therapy (dose >10mg/day prednisone or other equivocal hormone) has been discontinued for more than 2 weeks and who have no clinical evidence can be included;
3. Any previous treatment with PARP inhibitor, including, olaparib, niraparib, rucaparib, pamiparib, and fluzoparib;
4. Inability to swallow tablets properly or gastrointestinal function, may interfere with drug absorption, according to the investigator.
5. Recent (within 3 months) occurrence of intestinal obstruction, gastrointestinal perforation;
6. Patients with clinically symptomatic carcinomatous ascites or pleural effusion who need puncture or drainage or who have received drainage of ascites or pleural effusion within 2 months prior to the first trial of drug administration.
7. Patients with clinically significant cardiovascular disease that are not well controlled, such as (1) New York Heart Association (NYHA) ≥ grade 2 congestive heart failure (CHF) (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention (5) QTc > 470ms;
8. Patients with abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds), bleeding tendency, or who are receiving thrombolytic or anticoagulant therapy are permitted to receive low-dose low molecular heparin or oral aspirin for prophylactic anticoagulation during the trial;
9. Patients who have experienced clinically significant bleeding symptoms or have a definite bleeding tendency within 3 months prior to the first dose, such as peptic bleeding, bleeding gastric ulcer, or suffering from vasculitis, etc., may be retested if the fecal occult blood is positive at the baseline period, and if it is still positive after the retesting, combined with the clinical judgment, and if necessary, gastroscopy will be carried out;
10. Accompanied by active ulcers, unhealed wounds or with fractures;
11. Patients who suffering from hypertension which cannot be well controlled by antihypertensive medication (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 90mmHg);
12. Any bleeding event with a severity rating of 2 or more on the CTCAE 5.0 within 4 weeks prior to the first dose;
13. Patients has an active infection or an unexplained fever >38.5 degrees during the screening period, prior to the first dose;
14. Patients who has a congenital or acquired immune deficiency (e.g., HIV-infected), or active hepatitis (Hepatitis B reference: HBsAg-positive, HBV DNA ≥500 IU/ml; Hepatitis C reference: HCV antibody-positive, HCV viral copy number > upper limit of normal);
15. Prior history of radiotherapy, chemotherapy, hormonal therapy, or molecularly targeted therapy less than 4 weeks after completion of therapy (last dose) and prior to study drug administration (less than 5 drug half-lives for oral molecularly targeted agents); prior treatment-induced adverse events (other than alopecia) have not recovered to ≤ 1 degree (CTCAE 5.0);
16. Arterial/venous thrombotic events, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, occurred within 6 months prior to the first dose of medication.
17. Patients with an inherited or acquired history of bleeding or coagulation disorders (e.g. hemophiliacs, coagulation disorders, thrombocytopenia, etc.). There were clinically significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, etc., within 3 months prior to the first dose;
18. Patients has received other systemic antitumor therapy during the study period;
19. In the investigator's judgment, patients have other factors that may lead to the forced termination of the study, such as other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory test abnormalities, accompanied by family or social factors, which will affect the subject's safety, or the collection of information and samples.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-10-18 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | from the first drug administration up to 2 years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | from the first drug administration up to 5 years
  Time from the date of first study treatment administration to the date of death due to any cause.
Objective Response Rate (ORR) | from the first drug administration up to 2 years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time to start of first subsequent therapy or death (TFST) | from the first drug administration up to 5 years
  TFST is defined as the time from the first study administration to the earliest of the date of anti-cancer therapy start date following study treatment discontinuation, or death.
Time to start of second subsequent therapy or death (TSST) | from the first drug administration up to 5 years
  TSST is defined as the time from the first study administration to the earliest of the date of second subsequent anti-cancer therapy start date following study treatment discontinuation, or death.
Time to progression(TTP）by RECIST or CA-125 | from the first drug administration up to 5 years
  Time to progression by RECIST v. 1.1 or CA-125 or death is defined as the time from the first study administration to the date of RECIST or CA-125 progression or death by any cause, whichever occurs first.
Safety and tolerability | from the first drug administration up to 5 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
Patient Reported Outcomes (PROs) | from the first drug administration up to 5 years
  Determination of changes in PROs with EQ-5D-5L

OTHER OUTCOMES:
Exploratory endpoint | from the first drug administration up to 5 years
  Open collection of homologous recombination deficiency status (HRD) status was performed to assess the impact of HRD status on the efficacy of fluazoparib in combination with bevacizumab.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Cetntre, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided